CLINICAL TRIAL: NCT05444764
Title: PREdiCtIon of Weanability, Survival and Functional outcomEs After ECLS
Acronym: PRECISE - ECLS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Leiden University Medical Center (Other); Erasmus Medical Center (Other); St. Antonius Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Isala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dirk W. Donker, Prof. Dr., UMC Utrecht
Other Study IDs: 21-604
Record Dates: First submitted 2022-06-22; First posted 2022-07-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Extracorporeal Membrane Oxygenation; Extracorporeal Membrane Oxygenation Complication
Keywords: Extracorporeal life support; Extracorporeal membrane oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extracorporeal life support (ECLS) is used as a last resort intervention in patients with severe cardiac, circulatory and/or respiratory failure with high (>80%) expected mortality. Despite considerable improvements in patient selection and outcomes, mortality and morbidity after ECLS remain high. An improved selection and management of patients who are supported with ECLS is therefore unquestionably needed from a perspective of optimal patient care and the socio-economic impact of this costly intervention.

DETAILED DESCRIPTION:
This observational multicenter study was designed to serve the following objectives:

1. Develop a (dynamic) prediction tool for survival and quality of life outcomes 1 year after ECLS support for the situation at baseline and 7 days after ECLS initiation
2. Study the association between application of left ventricular unloading and ECLS support duration and weanability
3. Description of the incidence of VA ECLS weaning failure and identification of predictors for VA ECLS weaning failure

Under this umbrella research protocol, the data collected by this observational multicenter study can also be reused for potential novel substudies with the objective to improve the quality of care and the efficiency of current treatment strategies involving ECLS.

ELIGIBILITY:
Inclusion Criteria:

* Having received (VA and/or VV) ECLS
* All ECLS indications (refractory cardiac, circulatory and/or respiratory failure)
* Surgical and medical patients

Exclusion Criteria:

* < 18 years of age
* ECLS confined to cardiac surgery in the operating room (OR) or in the catheterization laboratory
* Objection against use of clinical data (opt-out principle)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ECLS patients treated at the UMCU (from 2012 onwards) and collaborating centers (May 2021 onwards) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
QoL | 1 year after admission
  By the EuroQol EQ-5D, an instrument to measure health related quality of life. It assesses health in five domains; mobility, self-care, usual activities, pain/discomfort and anxiety/depression, ranging from 1 to 3 in each domain (e.g. from 1 'I am not anxious or depressed' to 3 'I am extremely anxious or depressed' in the anxiety/depression domain) finding 243 unique health states. These health states can be converted into an index ranging from 0 (death) to 1 (perfect health)
Mortality | In-hospital mortality up to 30 days and through study completion, an average of 1 year.
Weaning success | In-hospital up to 30 days
  30 day survival without left ventricular assist device, heart transplantation or short Term mechanical support

SECONDARY OUTCOMES:
Complications | During ECLS support up to 30 days and 1 year
  Incidence of complications (infection, thrombosis, bleeding, respiratory and cardiovascular complications, mechanical complications, neurological complications)
ECLS support duration | ECLS days up to 30 days and 1 year
  Total duration (in days) of ECLS support
ICU admission length of stay | ICU days up to 30 days and 1 year
  Length of stay (in days) of ICU admission
30 day mortality | 30 days
60 day mortality | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Dirk W Donker, Professor, Principal Investigator — UMC Utrecht
Locations (6):
- Netherlands (6):
  - Catharinaziekenhuis Eindhoven, Eindhoven, North Brabant
  - Isala Hospital, Zwolle, Overijssel
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus Medisch Centrum, Rotterdam, South Holland
  - Antoniusziekenhuis Nieuwegein, Nieuwegein, Utrecht
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
Our data will be shared with third parties after approval of the Principle Investigator (in consideration with the participating centers). The criteria and time period will be determined on a case-by case basis.